CLINICAL TRIAL: NCT01570257
Title: A Randomized Trial of High and Low Pressure Level Settings on a Programmable Ventriculoperitoneal Shunt Valve for Idiopathic Normal Pressure Hydrocephalus. Results of the Dutch Evaluation Program Strata Shunt (DEPSS) Trial
Brief Title: A Trial of High and Low Pressure Level Settings on a Programmable Ventriculoperitoneal Shunt Valve for Idiopathic Normal Pressure Hydrocephalus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Isala (Other); Albert Schweitzer Hospital (Other); UMC Utrecht (Other); Atrium Medical Center (Other); University Medical Center Nijmegen (Other); Admiraal de Ruyter Hospital (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Ernst Delwel, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 03.1073
Record Dates: First submitted 2012-03-25; First posted 2012-04-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2012-03

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: normal pressure hydrocephalus; ventriculoperitoneal shunt; overdrainage; subdural effusion
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Subdural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): These patients receive a shunt with the valve preset and fixed at a Performance level of 1.0, corresponding to an opening/closing pressure of 35-55 mm H2O.
- Intervention group (Experimental): These patients receive a shunt with the valve preset at a Performance level (PL) of 2.5, corresponding to an opening/closing pressure of 135-155 mm H2O. The PL is allowed to be lowered until clinical improvement occurs.
  Interventions: Procedure: lowering of the performance level of an adjustable Strata valve in a ventriculoperitoneal (VP) shunt for treating idiopathic normal pressure hydrocephalus

INTERVENTIONS:
Procedure: lowering of the performance level of an adjustable Strata valve in a ventriculoperitoneal (VP) shunt for treating idiopathic normal pressure hydrocephalus — in the intervention group, the performance level(PL) of the valve of the VP shunt, preset at the highest PL (meaning highest resistance) is lowered stepwise in the follow-up period at 1,3 and 9 months postoperatively after implantation until improvement occurs or signs of overdrainage are encountered on a new CT scan of the brain. In the control group the PL is preset and fixed at the second lowest PL and these patients serve as a control group.
  Other Names: PS Medical Strata I valve (small) (Medtronic, Goleta, USA)
  Arms: Intervention group

SUMMARY:
In treating idiopathic normal pressure hydrocephalus with a shunt there is always a risk of underdrainage or overdrainage. The hypothesis is tested whether treatment of patients with an adjustable valve preset at the highest opening pressure (OPV), leads to comparable clinical results with less subdural effusions than in a control group with an opening pressure preset and kept fixed at a low pressure level.

DETAILED DESCRIPTION:
Idiopathic normal pressure hydrocephalus (INPH) is characterized by a clinical triad of symptoms: gait disturbance, urinary incontinence and cognitive impairment. INPH typically develops among the elderly and shares some symptoms with other neurological disorders. In general, 60-70% of patients with the complete clinical triad and signs of hydrocephalus on CT/MRI will improve after cerebrospinal fluid (CSF) shunting. Implantation of a shunt, however, carries complications such as infection, obstruction, underdrainage, and overdrainage. The cumulative complication rate and revision rate is estimated to be 35-80% among adults. The England shunt registry described an overall incidence of underdrainage of 52%, and studies have resulted in incidences of overdrainage between 2 and 21%. Børgesen claims that 80% of complications of shunting for INPH are related to overdrainage. Overdrainage may lead to low intracranial pressure syndrome and subdural effusions (SDE). Low intracranial pressure syndrome is characterized by orthostatic headaches and sometimes nausea, vomiting, drowsiness, diplopia, upward gaze palsy and visual defects. As INPH patients are often elderly patients with concomitant brain atrophy and normal CSF pressure they are especially at risk for developing signs and symptoms of overdrainage.

Overdrainage can be prevented or treated by implanting an anti-siphon device (ASD) or changing the opening pressure of the valve (OPV). Different ASDs have been developed since the first publication in 1973. They have in common that the lumen of the catheter is closed under influence of a negative hydrostatic pressure at the level of the ASD. The optimal valve setting for treating INPH is still the subject of controversy. The dilemma in INPH patients is that a low OPV might lead to overdrainage-related symptoms. A high valve setting might lead to underdrainage and the patient misses the chance of maximum improvement.

Studies examining whether to use a low or high OPV have been contradictory so far.

After randomization, baseline primary and secondary outcome measure assessments are conducted preoperatively. Within 24 hours of shunting, skull, thoracic, and abdominal X-rays are done to verify device connections and position. Follow-up visits at 1, 3, and 9 months include all primary and secondary outcome assessments. All measurements are done by a research assistant who visits the participating hospitals to prevent inter-observer variation. Study end for each patient is defined as completing the 9 month visit or death, detection of SDE on CT, or shunt removal or revision due to infection or dysfunction.

The PL in Group 1 (control group) is allowed to be increased to a higher setting when an SDE is detected. The patient thereby reaches study end, and the treating physician is free to decide how to manage the PL. The 9-month follow-up is still obtained. The PL in Group 2 is preset at the highest PL and eventually lowered 1 step at each follow-up visit when the modified mini mental state (3MS) or Gait score is not increased ≥ 15% provided that no SDE is visible on a new CT scan. The 15% is considered the minimum percentage to reliably determine improvement.

ELIGIBILITY:
Inclusion Criteria:

* At least two out of three of the typical signs of normal pressure hydrocephalus:

  * gait disturbance,
  * cognitive impairment and
  * urinary incontinence.
* Radiological verification of a communicating hydrocephalus.
* Cerebrospinal fluid pressure at lumbar puncture < 150 mm H2O.

Exclusion Criteria:

* Aqueduct stenosis.
* Severe comorbidity.
* Age > 85 years.
* Possibly confounding neurological diseases.
* Recent meningitis or subarachnoid hemorrhage.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-09; Primary Completion 2006-12 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
the number of Subdural effusions, detected on CT scan, in patients showing clinical improvement after implantation of a ventriculoperitoneal shunt,at the end of the study | baseline and 9 months (end of study)
  the most important parameter of the study will be the difference in incidence of subdural effusions between both groups

SECONDARY OUTCOMES:
the final performance level of the valve of the shunt at the end of the study | baseline and 9 months (end of study)
  Peformance level is the opening/closing pressure of the valve and reflects the hydrostatic resistance of the valve of the shunt
change in gait score | baseline and 9 months (end of study)
change in urinary incontinence | baseline and 9 months (end of study)
change in modified mini mental state (3MS) score | baseline and 9 months (end of study)
  the 3MS score quantifies cognitive function
change in modified Rankin (mRS) score | baseline and 9 months (end of study)
  the mRS quantifies functional impairment
change in Evans' ratio | baseline and 9 months (end of study)
  a measure of ventricular width, on CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Clemens MF Dirven, Prof. PhD, Study Chair — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands